CLINICAL TRIAL: NCT05420831
Title: Comparison the Effectiveness and Safety of Vaginal and Laparoscopic Apical Fixation Techniques Using a Synthetic Mesh for Pelvic Organ Prolapse Treatment. A Randomized Controlled Study
Brief Title: Comparison of Vaginal and Laparoscopic Apical Fixation Techniques for Pelvic Organ Prolapse Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Shkarupa Dmitry, Ph.D., Deputy Director for medical care, Chief Urologist of Saint Petersburg State University Clinic of advanced medical technologies n.a. N.I.Pirogov., Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vaginal_or_laparoscopic
Record Dates: First submitted 2022-05-18; First posted 2022-06-15 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: sacrohysteropexy; pelvic organ prolapse; apical prolapse; vaginal repair; vaginal mesh; sacrospinous fixation
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacrospinous fixation of the vaginal apex with the synthetic mesh (Active Comparator)
  Interventions: Procedure: Vaginal
- Laparoscopic sacrocolpopexy (Active Comparator)
  Interventions: Procedure: Laparoscopic

INTERVENTIONS:
Procedure: Vaginal — Sacrospinous hysteropexy using the synthetic mesh
  Arms: Sacrospinous fixation of the vaginal apex with the synthetic mesh
Procedure: Laparoscopic — Laparoscopic Sacrohysteropexy
  Arms: Laparoscopic sacrocolpopexy

SUMMARY:
This is a prospective randomized controlled study, designed to compare efficacy and safety of two methods of apical fixation in patients with pelvic organ prolapse (POP) - sacrospinous hysteropexy (SSHP) with synthetic mesh and laparoscopic sacrohysteropexy (LSHP), and the impact of the surgery on quality of life.

DETAILED DESCRIPTION:
BACKGROUND POP remains a widespread condition, that significantly affects patients' quality of life. The estimated incidence of POP in women varies from 10% in young age to 40% after menopause. Apical defect is the least frequent of all types of POP and occurs in 5-15% of patients, however apical support is crucial to maintaining normal anatomy of the pelvic floor.

Although the uterus itself is not the cause of POP, hysterectomy is the most common surgery for POP. However there is a growing interest in uterine-sparing surgical techniques because a lot of women express a desire to preserve uterus.

There are various techniques for uterine-sparing apical repair, including abdominal (laparoscopic or robotic) and vaginal apical fixation. SSHP is the most studied method of apical fixation and was originally performed with sutures. The use of transvaginal mesh for SSHP is discussable in conjunction with numerous reports of complications and wariness towards synthetic materials use. Some authors though reported of comparable effectiveness and high safety of SSHP using mesh. Due to the lack of the reliable evidence, to date there are no consensus about optimal method of hysteropexy, as LSHP is not without its drawbacks and complications.

PREOPERATIVE ASSESSMENT All patients who meet eligibility criteria will undergo a preoperative assessment: medical history, physical and vaginal examination, assessing pelvic organ prolapse according to Pelvic Organ Prolapse Quantification System (POP-Q). All patients will complete questionnaires validated in Russia: Pelvic Floor Disability Index (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire, short form (PISQ-SF), Patient Global Impression of Improvement (PGI-I).

MATERIALS AND METHODS The investigators hypothesis is that SSHP is non-inferior to LSHP in terms of recurrence rate and complications. The sample size was calculated assuming an objective cure rate of 92% as described in literature. With a power of 80%, a level of 0,05 and the non-inferiority margin at 15%, the sample size is 92 patients. The investigators assume a drop-out rate of 10%, thus a total of 102 participants will be included in the study.

All enrolled patients will be randomly assigned to SSHP or LSHP treatment groups in equal ratio the day before the surgery, using computer randomization.

All data will be collected by medical staff not involved in treatment. Collected pre- and postoperative data will be anonymized using unique codes, that patients will receive immediately after randomization.

All surgical interventions will be performed by 3 qualified surgeons. Postoperative follow-up will be performed 6, 12 and 24 months after surgery by 2 researchers, who will be blinded about the type of intervention.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a woman with anterior and apical compartment pelvic organ prolapse
* The age of a subject is 45-80 years
* Leading point of prolapse is at the level of the hymen or distal to the hymen (Ba, C>=0 according to POP-Q classification)
* The subject gave written consent to participate in the study
* The subject is able to evaluate the risks of the treatment and make an independent decision on participation in the study
* The subject is able to fill up validated questionnaires and come to the control visit after the surgery

Exclusion Criteria:

* The subject has an active urinary tract infection or skin infection in the region of surgery or acute infectious disease
* The subject had prior surgery for POP, stress urinary incontinence (SUI) or hysterectomy
* The subject has history of pelvic cancer
* The subject has chronic pelvic pain
* The subject has cervical elongation
* The subject has severe obesity (BMI > 30)
* The subject has postoperative scars/suspected adhesions in the ares of surgical access to the abdomen
* The subject has gynecological diseases (recurrent uterine bleeding, endometrial hyperplasia, the presence of atypical cells in cervical smears, adenomyosis, multiple uterine myoma)
* The subject has urinary incontinence
* The subject is planning pregnancy
* The subject is unable to visit postoperative check-ups
* Refusal from participation.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
Objective cure rate | 24 months (2 years)
  The patient is considered cured if there is no prolapse beyond the hymen and the cervix is above -1 cm according to POP-Q (0-1 stage)

SECONDARY OUTCOMES:
Satisfaction with the surgery | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Measured through the Patient Global Impression of Improvement questionnaire (PGI-I), validated in Russia. The patient marks the number that best describes her post-operative condition, compared with how it was before surgery. The score ranges from 1 (very much better) to 7 (very much worse).
The impact of treatment on sexual function | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Measured through the scoring of Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) validated in Russia. The scale evaluates sexual function in patients with urinary incontinence and/or POP. The responses are graded on a five-point Likert scale ranging from 0 (always) to 4 (never). Items 1 - 4 are reversely scored and a total of 48 is the maximum score. The higher scores indicate better sexual function.
The impact of treatment on the quality of life | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Measured through the Pelvic Floor Disability Index (PFDI-20), validated in Russia. The item includes 20 questions. The score ranges from 0 to 300. The higher the score, the worse the outcome.
Observed complications | Measured postoperatively at intervals of 6, 12 and 24 months postoperatively
  Presence of any adverse effects such as: bleeding requiring blood transfusion, haematoma, organ perforation, nerve injury, vaginal scarring and shortening, wound infection, urinary tract infection, pelvic pain, mesh extrusion in the vagina, mesh erosion into the urinary tract, dyspareunia de novo, de novo urgency, atonic bladder, de novo stress urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Shkarupa, MD, PhD, Study Chair — Saint Petersburg State University, Russia
Locations (1):
- Saint-Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No